CLINICAL TRIAL: NCT03766698
Title: Muscle Architecture of Lower Extremity In Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, zekiye ipek katırcı kırmacı, Principal Investigator, Sanko University
Other Study IDs: SankoUniversity
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Muscle Architecture; Lower extremity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to determine the muscle architecture of the lower extremity muscles (pennation angle, muscle fiber length and muscle thickness) in patients with multiple sclerosis. Lower extremity muscles of patients with multiple sclerosis and healthy individuals; rectus femoris, biceps femoris, tibialis anterior, gastrosoleus and gastrocnemius muscles will be examined by ultrasound method.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is characterised by complex and heterogeneous symptoms, often leading to reduced quality of life and impaired functional capacity. The latter is related to reduced muscle strength of predominately the lower limbs . The mechanisms underlying the observed strength deficits are of muscular as well as neural origin . At the whole muscle level, a number of studies have examined skeletal muscle characteristics of MS patients, with some studies but not all, reporting loss of muscle mass and decreased or comparable maximal muscle strength.

However, there is no study describing the features of lower extremity muscle architecture in multiple sclerosis. Muscle architecture is defined as the alignment of muscle fibers with respect to the axis of force. Although the diameters of the muscles of different sizes are quite similar to the diameters of the fibers, the sequences of these fibers contain several differences. The alignment of the muscle forming fibers has a significant effect on the force of muscle formation. The parameters that determine muscle architecture characteristics are the muscle fiber length, pennation angle, the physiological cross-sectional area. For each muscle these parameters may differ from each other. Any type of load in the case is the result of an adaptation process that results in muscle development. Muscle architecture allows the macroscopic understanding and interpretation of this adaptation process.

Determining the muscle architecture of multiple sclerosis patients by ultrasound will guide the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Individuals who agree to be voluntary,
* With the EDSS 4 and below
* Without pregnancy
* Do not receive corticosteroid treatment in the last month
* Do not take any medicine that will affect walking in the last 1 month

Exclusion Criteria:

* Those who refuse to volunteer,
* EDSS over 4
* Pregnancy
* Corticosteroid therapy within 1 month
* Any medication that will affect walking in the last 1 month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study Population consists of Multiple Sclerosis Patients and Healthy Volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Muscle Architecture Pennation Angle | The evaluation will be made on the first 1 day.
  Pennation Angle will be assesed by ultrasound imaging.
Muscle Architecture Muscle Fiber Lengh | The evaluation will be made on the first 1 day.
  Muscle Fiber Lenght will be assesed by ultrasound imaging.
Muscle Architecture Muscle Thickness | The evaluation will be made on the first 1 day.
  Muscle Thickness will be assesed by ultrasound imaging.

SECONDARY OUTCOMES:
Muscle Strength | The evaluation will be made on the first 1 day.
  Ouadriceps, Hamstring, Gastrosoleus and Gastrocnemius muscle Strenght will be asses with digital hand-held dynamometer (Commander PowerTrack II muscle tester).
Circumference Measurement of Thigh | The evaluation will be made on the first 1 day.
  Thigh circumference will be measured with a tape measure. Thigh circumference measurement will be measured from the midline of the inguinal line and superior patella.
Circumference Measurement of shin | The evaluation will be made on the first 1 day.
  Shin circumference will be measured with a tape measure.Shin circumference measurement will be measured from the poplital line and the middle point of the achilles.

OTHER OUTCOMES:
Thickness of subcutaneous fat from anterior thigh | The evaluation will be made on the first 1 day.
  Subcutaneous fat will be assesed with skinfold from anterior thigh. At the same time the thickness of subcutaneous fat will also be evaluated by ultrasound imaging.
Thickness of subcutaneous fat from posterior leg | The evaluation will be made on the first 1 day.
  Subcutaneous fat will be assesed with skinfold from posterior leg. At the same time the thickness of subcutaneous fat will also be evaluated by ultrasound imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Sanko University
Locations (1):
- Sanko University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of data information has not yet been decided.

REFERENCES:
- [Result] Wens I, Dalgas U, Vandenabeele F, Krekels M, Grevendonk L, Eijnde BO. Multiple sclerosis affects skeletal muscle characteristics. PLoS One. 2014 Sep 29;9(9):e108158. doi: 10.1371/journal.pone.0108158. eCollection 2014. PMID 25264868
- [Derived] Kirmaci ZIK, Firat T, Ozkur HA, Neyal AM, Neyal A, Ergun N. Muscle architecture and its relationship with lower extremity muscle strength in multiple sclerosis. Acta Neurol Belg. 2022 Dec;122(6):1521-1528. doi: 10.1007/s13760-021-01768-1. Epub 2021 Aug 20. PMID 34417688
- See also: Multiple Sclerosis and Skeletal Muscle — https://www.ncbi.nlm.nih.gov/pubmed/25264868